CLINICAL TRIAL: NCT01857362
Title: A Study to Evaluate the Bioequivalence of Orfadin Capsules 20 mg Compared to Orfadin Capsules 10 mg. An Open-label, Randomized, Cross-over, Single-dose Study in Healthy Volunteers.
Brief Title: Bioequivalence of Orfadin 20 mg Compared to Orfadin 10 mg Capsules.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Sobi.NTBC-004
Record Dates: First submitted 2013-05-16; First posted 2013-05-20 (Estimated); Results first posted 2014-10-27 (Estimated); Last update posted 2021-10-12 (Actual); Status verified 2021-09

CONDITIONS: Healthy
Keywords: Orfadin; Nitisinone; Bioequivalence
MeSH Terms: interventions — nitisinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nitisinone 2 x 10 mg (Active Comparator): Two nitisinone 10 mg capsules by mouth as a single dose
  Interventions: Drug: Nitisinone 10 mg
- Nitisinone 1 x 20 mg capsule (Experimental): One nitisinone 20 mg capsule by mouth as a single dose
  Interventions: Drug: Nitisinone 20 mg

INTERVENTIONS:
Drug: Nitisinone 20 mg — Nitisinone 20 mg capsules
  Arms: Nitisinone 1 x 20 mg capsule
Drug: Nitisinone 10 mg — Nitisinone 10 mg capsules
  Arms: Nitisinone 2 x 10 mg

SUMMARY:
The purpose of this study is to evaluate the bioequivalence between Orfadin 20 mg and 10 mg capsules in healthy volunteers.

DETAILED DESCRIPTION:
This is an open, randomized 2-way crossover study in 12 healthy volunteers. Subjects will receive single oral 20 mg doses of nitisinone administrated as one 20 mg capsule or as two 10 mg capsules of Orfadin. There will be a 3-week washout period between the doses.

There will be a screening visit within 3 weeks prior to the first dose. During each treatment period, subjects will be admitted to the clinic from the afternoon on the day before drug administration (i.e., on Day -1) and remain at the clinic until the 48-hour post-dose blood sample has been collected in the morning of Day 3. They will then return for ambulatory visit in the morning of Day 4 (72-hour sample). A follow-up visit will take place 7-14 days after the last dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers between 18-55 years of age, inclusive.
* BMI between 18,5-30,0 kg/m2, inclusive.

Exclusion Criteria:

* Subjects with current keratopathy, or other abnormalities found by slit-lamp examination.
* Subjects who are heavy smokers or consume more than 5 cups of coffee per day.
* Subjects with history of drug and/or alcohol abuse or a positive drug screen or alcohol breath test.
* Subjects with positive screens for hepatitis B surface antigen, hepatitis C antibodies and human immunodeficiency virus (HIV) 1-2 antibodies.
* Subjects who were enrolled in another concurrent clinical study or intake of an investigational medicinal product within three months prior to inclusion in this study.
* Subjects who donate more than 50 mL of blood within 60 days prior to drug administration or donate more than 1,5 liters of blood in the 10 months prior to first drug administration.
* Female subjects that are pregnant or breastfeeding.
* Female subjects of childbearing potential and all male subjects must be willing to use effective forms of contraception.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erik Brouwer, MD, Study Director — Swedish Orphan Biovitrum
Locations (1):
- Pharmaceutical Research Associates Group B.V (PRA), Zuidlaren, Netherlands

RESULTS

PARTICIPANT FLOW:
Groups:
- Nitisinone 1 x 20 mg, Then Nitisinone 2 x 10 mg: Participants first received one nitisinone capsule of 20 mg. After washout of 3 weeks participants then received two nitisinone capsules of 10 mg.
- Nitisinone 2 x 10 mg, Then Nitisinone 1 x 20 mg: Participants first received two nitisinone capsules of 10 mg. After washout of 3 weeks participants then received one nitisinone capsule of 20 mg.
Period: Overall Study
Arm/Group | Nitisinone 1 x 20 mg, Then Nitisinone 2 x 10 mg | Nitisinone 2 x 10 mg, Then Nitisinone 1 x 20 mg
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: All treatment arms
Arm/Group | Overall Study
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (11)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Region of Enrollment [Number; unit: participants]
  Netherlands | 12

OUTCOME MEASURES:

1. Primary Outcome: The Area Under the Serum Concentration vs. Time Profile During 72 Hours After Dose (AUC72h).
Time Frame: Day 1 predose and at 15, 30, 45 minutes and 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours postdose
Population: Full analysis set was used; subjects with available PK data for at least one of the treatments.
Measure: Geometric Mean (Full Range); unit: uM*h
Groups:
- Nitisinone 2 x 10 mg Capsules: Nitisinone 2 x 10 mg capsules
- Nitisinone 1 x 20 mg Capsules: Nitisinone 1 x 20 mg capsules
Arm/Group | Nitisinone 2 x 10 mg Capsules | Nitisinone 1 x 20 mg Capsules
Number analyzed (Participants) | 12 | 12
uM*h | 262 [209 to 336] | 267 [210 to 341]
Statistical Analysis 1: Comparison: Nitisinone 2 x 10 mg Capsules vs Nitisinone 1 x 20 mg Capsules; Test type: Non-Inferiority or Equivalence — Bioequivalence is established if the 90% confidence interval for the ratio is completely within the acceptance range (0.80-1.25); ANOVA; Ratio of geomectric means = 1,016, 90% CI 2-sided [0.988 to 1.045]

2. Primary Outcome: The Maximum Serum Concentration (Cmax).
Time Frame: Day 1 predose and at 15, 30, 45 minutes and 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours postdose
Population: Full analysis set was used; subjects with available PK data for at least one of the treatments.
Measure: Geometric Mean (Full Range); unit: nM
Arm/Group | Nitisinone 2 x 10 mg Capsules | Nitisinone 1 x 20 mg Capsules
Number analyzed (Participants) | 12 | 12
nM | 6438 [4510 to 8950] | 6366 [4690 to 9330]
Statistical Analysis 1: Comparison: Nitisinone 2 x 10 mg Capsules vs Nitisinone 1 x 20 mg Capsules; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; ratio of geometric means = 0.989, 90% CI 2-sided [0.945 to 1.034]

ADVERSE EVENTS:
Arm/Group | Nitisinone 2 x 10 mg Capsules | Nitisinone 1 x 20 mg Capsules
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 4/12 | 4/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nitisinone 2 x 10 mg Capsules (N=12) | Nitisinone 1 x 20 mg Capsules (N=12)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Catheter site related reaction (General disorders) | 0 (0) | 1 (1)
Hunger (General disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days